CLINICAL TRIAL: NCT00295841
Title: A Phase I Open-Label Study of High-Dose Cytarabine and Clofarabine in Adult Patients With Refractory or Relapsed Acute Myelogenous Leukemia or Refractory or Relapsed Acute Lymphoblastic Leukemia
Brief Title: Cytarabine and Clofarabine in Treating Patients With Refractory or Relapsed Acute Myeloid Leukemia or Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000466307; CCCWFU-21204; ILEX-CCCWFU-21204; CCCWFU-BG04-519
Record Dates: First submitted 2006-02-23; First posted 2006-02-24 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Leukemia
Keywords: recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute basophilic leukemia; adult acute eosinophilic leukemia; adult erythroleukemia (M6a); adult pure erythroid leukemia (M6b); adult acute megakaryoblastic leukemia (M7); adult acute minimally differentiated myeloid leukemia (M0); adult acute monoblastic leukemia (M5a); adult acute monocytic leukemia (M5b); adult acute myeloblastic leukemia with maturation (M2); adult acute myeloblastic leukemia without maturation (M1); adult acute myelomonocytic leukemia (M4)
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Basophilic, Acute; Leukemia, Eosinophilic, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myelomonocytic, Acute | interventions — Clofarabine; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: clofarabine
Drug: cytarabine

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cytarabine and clofarabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells.

PURPOSE: This phase I trial is studying the side effects and best dose of clofarabine when given together with cytarabine and to see how well they work in treating patients with refractory or relapsed acute myeloid leukemia or acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate in adult patients with relapsed or refractory acute myeloid leukemia or acute lymphoblastic leukemia treated with high-dose cytarabine followed by clofarabine.
* Document the safety profile and tolerability of this regimen in these patients.
* Phase I: Patients receive high-dose cytarabine IV over 3 hours followed by clofarabine IV over 2 hours on days 1-5. Treatment repeats for up to 4 courses (1-2 induction courses, 2-3 post-remission courses) in the absence of disease progression or unacceptable toxicity.

A cohort of 3-6 patients receives the starting dose of clofarabine. If 1 of 6 patients experiences dose-limiting toxicity (DLT), a subsequent cohort of patients receives clofarabine at the next higher dose. If ≥ 2 of 6 patients experience DLT, the dose of cytarabine is reduced and subsequent cohorts of patients receive cytarabine at reduced doses and clofarabine as per the dose-escalation scheme above.

PROJECTED ACCRUAL: A total of 9 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Pathologic confirmation of acute myeloid leukemia (AML) or acute lymphoblastic leukemia (ALL)

  * No M3 AML
* Meets 1 of the following criteria:

  * In first relapse
  * In second relapse after a second complete remission (CR) that lasted ≥ 3 months
  * Refractory to initial induction therapy
* No symptomatic CNS involvement

PATIENT CHARACTERISTICS:

* ECOG performance status ≤ 2
* Creatinine < 2 mg/dL
* Bilirubin ≤ 2 mg/dL
* AST and ALT ≤ 4 times upper limit of normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 2 weeks after completing study treatment
* Ejection fraction ≥ 45% by echocardiogram
* No active, uncontrolled systemic infection considered opportunistic, life-threatening, or clinically significant
* No psychiatric disorders that would interfere with giving consent, study participation, or follow-up procedures
* No other severe concurrent disease that would preclude study treatment

PRIOR CONCURRENT THERAPY:

* At least 1 week since prior therapy and recovered
* No other concurrent chemotherapy

  * Hydroxyurea to control WBC count before starting study treatment allowed
* No concurrent corticosteroids unless used for diseases other than leukemia
* No concurrent palliative radiotherapy
* No concurrent growth factors (e.g., epoetin alfa, filgrastim [G-CSF], or sargramostim [GM-CSF]) in patients with AML

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2005-02; Primary Completion 2015-01-07 (Actual); Study Completion 2015-01-07 (Actual)

PRIMARY OUTCOMES:
Response rate
Safety profile and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Bayard L. Powell, MD, Study Chair — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina, United States